CLINICAL TRIAL: NCT02565732
Title: Safety and Efficacy of Botulinum Toxin Type A Topical Gel for Primary Axillary Hyperhidrosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Revance Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RT001-CL045
Record Dates: First submitted 2015-09-29; First posted 2015-10-01 (Estimated); Last update posted 2016-08-04 (Estimated); Status verified 2016-03

CONDITIONS: Hyperhidrosis
MeSH Terms: conditions — Hyperhidrosis | interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- Dose A (Experimental): Botulinum toxin type A
  Interventions: Biological: Botulinum toxin type A
- Dose B (Experimental): Botulinum toxin type A
  Interventions: Biological: Botulinum toxin type A
- Dose C (Placebo Comparator): Placebo comparator
  Interventions: Biological: Placebo comparator

INTERVENTIONS:
Biological: Botulinum toxin type A — Botulinum toxin type A, Dose A, Topical
  Arms: Dose A
Biological: Botulinum toxin type A — Botulinum toxin type A, Dose B, Topical
  Arms: Dose B
Biological: Placebo comparator — Placebo, Dose C, Topical
  Arms: Dose C

SUMMARY:
This is a safety and efficacy study of botulinum toxin type A in subjects with primary axillary hyperhidrosis.

ELIGIBILITY:
Inclusion Criteria:

* Primary axillary hyperhidrosis
* Female or male, 18 years of age or older in good general health
* Excessive sweating interferes with daily life activities and scores 3 or 4 on the HDSS at Screening and Baseline
* Axillary sweat production of at least 50 mg/5 min measured gravimetrically

Exclusion Criteria:

* Any neurological condition, that may place the subject at increased risk with exposure to botulinum toxin type A such as amyotrophic lateral sclerosis and motor neuropathy, Lambert-Eaton syndrome, and Myasthenia gravis
* Muscle weakness or paralysis, particularly in the upper extremities
* Active skin disease or irritation or disrupted barrier at the treatment area
* Undergone any procedures which may affect the axillary areas
* Treatment with botulinum toxin type A in the axilla in the last 9 months or anywhere in the body in the last 6 months
* Any prior axillary use of an anti-hyperhidrosis medical device
* If menopausal had symptoms of menopause such as sweating or flushing within the last year

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2015-09; Primary Completion 2015-12 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Hyperhidrosis Disease Severity Scale (HDSS) | Week 4
  Improvement at follow-up in the experimental groups compared to the placebo group
Gravimetry | Week 4
  The amount of sweat measured gravimetrically

SECONDARY OUTCOMES:
Dermatology Life Quality Index (DLQI) | Week 4

CONTACTS AND LOCATIONS:
Locations (1):
- San Francisco, California, United States